CLINICAL TRIAL: NCT03078582
Title: Phase 2 Multicenter, Open-Label, Uncontrolled Study to Evaluate the Safety, Tolerability, Efficacy, Pharmacokinetics, and Pharmacodynamics of RA101495 in Subjects With Paroxysmal Nocturnal Hemoglobinuria
Brief Title: Phase 2 Safety and Efficacy Study of Zilucoplan (RA101495) to Treat PNH Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ra Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RA101495-01.201; 2016-003522-16 (EudraCT Number)
Record Dates: First submitted 2017-03-08; First posted 2017-03-13 (Actual); Results first posted 2020-03-10 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
Keywords: PNH
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — zilucoplan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zilucoplan (RA101495) treatment naive (Experimental): 0.3mg/kg subcutaneously (SC) at Day 1 (loading dose) followed by a starting maintenance dose of 0.1 mg/kg daily SC (treatment naïve)
  Interventions: Drug: Zilucoplan (RA101495)
- Zilucoplan (RA101495) previously on eculizumab (Experimental): 0.3mg/kg subcutaneously (SC) at Day 1 (loading dose) followed by a starting maintenance dose of 0.1 mg/kg daily SC (previously on eculizumab)
  Interventions: Drug: Zilucoplan (RA101495)

INTERVENTIONS:
Drug: Zilucoplan (RA101495) — 0.3mg/kg subcutaneously (SC) at Day 1 (loading dose) followed by a starting maintenance dose of 0.1 mg/kg daily SC

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of zilucoplan (RA101495) in patients with Paroxysmal Nocturnal Hemoglobinuria (PNH). There will be two groups of patients in the study: the first group will include patients who have never received eculizumab for treatment of PNH. The second group will include patients who have received treatment with eculizumab for at least 6 months prior to the study. Patients will be treated with RA101495 for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PNH by flow cytometry
* For treatment naive patients: subjects must not have received treatment with eculizumab prior to or during the Screening Period and must have a lactate dehydrogenase (LDH) level ≥2 times the upper limit of normal (xULN) during Screening
* For patients who previously received eculizumab: subjects must have received treatment with eculizumab for at least 6 months prior to Screening

Exclusion Criteria:

* History of meningococcal disease
* Current systemic infection or suspicion of active bacterial infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Anita Hill, Principal Investigator — St James' Institute of Oncology
Locations (12):
- Australia (2):
  - Investigative Site, Gosford, New South Wales
  - Investigative Site, Parkville
- Investigative Site, Toronto, Ontario, Canada
- Investigative Site, Copenhagen, Denmark
- Investigative Site, Helsinki, Finland
- Germany (2):
  - Investigative Site, Essen
  - Investigative Site, Ulm
- Investigative Site, Budapest, Hungary
- New Zealand (2):
  - Investigative Site, Christchurch
  - Investigative Site, Hamilton
- United Kingdom (2):
  - Investigative Site, Leeds
  - Investigative Site, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://learningcenter.ehaweb.org/eha/2018/stockholm/214782/anita.hill.ra101495.a.subcutaneously-administered.peptide.inhibitor.of.html?f=menu=14*media=3*speaker=664274

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A (Treatment Naive); Cohort B (Previously on Eculizumab): 0.3mg/kg subcutaneously (SC) at Day 1 (loading dose) followed by a starting maintenance dose of 0.1 mg/kg daily SC
Period: Overall Study
Arm/Group | Cohort A (Treatment Naive) | Cohort B (Previously on Eculizumab)
Started | 10 | 16
Completed | 10 | 8
Not Completed | 0 | 8
Not completed — Adverse Event | 0 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A (Treatment Naive) | Cohort B (Previously on Eculizumab) | Total
Number analyzed (Participants) | 10 | 16 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 11 | 18
  >=65 years | 3 | 5 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (14.5) | 49.6 (18.5) | 53.4 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 4 | 9 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 10 | 14 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  New Zealand | 4 | 0 | 4
  Canada | 1 | 0 | 1
  Hungary | 1 | 1 | 2
  Finland | 1 | 2 | 3
  Denmark | 0 | 1 | 1
  United Kingdom | 2 | 3 | 5
  Australia | 0 | 5 | 5
  Germany | 1 | 4 | 5
Weight [Mean (Standard Deviation); unit: kg] | 77.77 (20.64) | 79.16 (14.86) | 78.63 (16.92)
Height [Mean (Standard Deviation); unit: cm] | 168.25 (11.08) | 171.10 (8.69) | 170.00 (9.56)
BMI [Mean (Standard Deviation); unit: kg/m2] | 27.30 (6.15) | 26.95 (4.14) | 27.08 (4.89)

OUTCOME MEASURES:

1. Primary Outcome: Change-from-baseline in Serum Lactate Dehydrogenase (LDH) Level.
Description: The primary efficacy endpoint is the change-from-baseline in serum LDH levels during this period, defined as the mean LDH values of Weeks 6, 8, 10, and 12 minus the baseline value of LDH.
Time Frame: Through Week 12 of the study
Population: Efficacy Evaluable
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Cohort A (Treatment Naive) | Cohort B (Previously on Eculizumab)
Number analyzed (Participants) | 10 | 8
U/L | -695.2 (589.2) | 216.7 (209.2)

2. Secondary Outcome: Changes From Baseline in Bilirubin Values
Description: Changes from baseline at each of the scheduled post-baseline time-points
Time Frame: Through Week 12 of the study
Population: Efficacy Evaluable
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Cohort A (Treatment Naive) | Cohort B (Previously on Eculizumab)
Number analyzed (Participants) | 10 | 8
umol/L
  Week 1: number analyzed (Participants) | 10 | 7
  Week 1 | 1.3 (7.2) | 1.9 (4.5)
  Week 2 | 3.1 (7.7) | 4.4 (6.5)
  Week 3 | 4.4 (9.0) | 6.8 (7.5)
  Week 4 | 4.0 (6.7) | 4.3 (6.5)
  Week 6 | 4.1 (7.4) | 3.8 (7.8)
  Week 8 | 4.0 (6.1) | 4.4 (9.9)
  Week 10 | 5.7 (10.9) | 1.5 (6.1)
  Week 12 | 4.6 (11.8) | 0.9 (4.5)

3. Secondary Outcome: Total Hemoglobin
Description: Changes from baseline at each of the scheduled post-baseline time-points
Time Frame: Through Week 12 of the Study
Population: Efficacy Evaluable
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Cohort A (Treatment Naive) | Cohort B (Previously on Eculizumab)
Number analyzed (Participants) | 10 | 8
g/L
  Week 1: number analyzed (Participants) | 10 | 7
  Week 1 | -1.5 (10.4) | -0.7 (7.1)
  Week 2 | 1.6 (7.4) | 0.9 (5.4)
  Week 3 | 4.3 (9.5) | -1.1 (9.0)
  Week 4 | 2.7 (10.5) | -0.9 (5.1)
  Week 6 | 3.6 (9.8) | -1.4 (5.3)
  Week 8 | 3.1 (9.6) | -1.0 (7.6)
  Week 10 | 4.5 (8.8) | -1.3 (8.7)
  Week 12 | 6.9 (10.6) | 0.5 (7.2)

4. Secondary Outcome: Changes From Baseline in Free Hemoglobin Values
Description: Changes from baseline at each of the scheduled post-baseline time-points
Time Frame: Through Week 12 of the study
Population: Efficacy Evaluable
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cohort A (Treatment Naive) | Cohort B (Previously on Eculizumab)
Number analyzed (Participants) | 10 | 8
mg/dL
  Week 1: number analyzed (Participants) | 8 | 8
  Week 1 | -7.84 (8.37) | 3.55 (18.51)
  Week 2: number analyzed (Participants) | 9 | 8
  Week 2 | -8.31 (9.07) | -1.00 (11.66)
  Week 3: number analyzed (Participants) | 8 | 8
  Week 3 | -5.65 (10.25) | -0.21 (3.87)
  Week 4: number analyzed (Participants) | 9 | 8
  Week 4 | -7.57 (8.12) | 16.90 (50.64)
  Week 6: number analyzed (Participants) | 8 | 7
  Week 6 | -8.24 (9.19) | -3.53 (10.66)
  Week 8: number analyzed (Participants) | 9 | 8
  Week 8 | -7.62 (9.07) | -2.39 (9.25)
  Week 10: number analyzed (Participants) | 9 | 8
  Week 10 | -7.60 (9.03) | -2.02 (10.06)
  Week 12: number analyzed (Participants) | 8 | 7
  Week 12 | -7.39 (10.10) | -2.23 (11.32)

5. Secondary Outcome: Haptoglobin Values
Description: Changes from baseline at each of the scheduled post-baseline time-points
Time Frame: Through Week 12 of the Study
Population: Efficacy Evaluable
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Cohort A (Treatment Naive) | Cohort B (Previously on Eculizumab)
Number analyzed (Participants) | 10 | 8
g/L
  Week 1 | 0.090 (0.285) | 0.010 (0.019)
  Week 2 | 0.080 (0.253) | -0.003 (0.007)
  Week 3 | 0.006 (0.019) | -0.003 (0.007)
  Week 4 | 0.012 (0.038) | -0.064 (0.180)
  Week 6 | 0.000 (0.000) | -0.064 (0.180)
  Week 8 | 0.004 (0.013) | -0.064 (0.180)
  Week 10 | 0.000 (0.000) | -0.064 (0.180)
  Week 12 | 0.000 (0.000) | -0.064 (0.180)

6. Secondary Outcome: Reticulocyte Values
Description: Changes from baseline at each of the scheduled post-baseline time-points
Time Frame: Through Week 12 of the Study
Population: Efficacy Evaluable
Measure: Mean (Standard Deviation); unit: 10^12 cells/L (SI Units)
Arm/Group | Cohort A (Treatment Naive) | Cohort B (Previously on Eculizumab)
Number analyzed (Participants) | 10 | 8
10^12 cells/L (SI Units)
  Week 1: number analyzed (Participants) | 10 | 7
  Week 1 | -0.0113 (0.0494) | -0.0147 (0.0326)
  Week 2 | -0.0157 (0.0591) | 0.0022 (0.0279)
  Week 3 | -0.0099 (0.0584) | 0.0063 (0.0197)
  Week 4 | -0.0137 (0.0439) | 0.0004 (0.0289)
  Week 6 | 0.0000 (0.0538) | 0.0170 (0.0259)
  Week 8 | -0.0042 (0.0619) | 0.0050 (0.0346)
  Week 10 | -0.0060 (0.0608) | 0.0085 (0.0304)
  Week 12 | -0.0047 (0.0570) | 0.0061 (0.0166)

7. Secondary Outcome: Hemoglobinuria Values
Description: Changes from baseline at each of the scheduled post-baseline time-points; Hemoglobinuria was assessed using a urine colorimetric scoring system with a score of 1 through 10. Where 1 represents no hemoglobinuria and 10 represents maximum hemoglobinuria.
Time Frame: Through Week 12 of the Study
Population: Efficacy Evaluable
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort A (Treatment Naive) | Cohort B (Previously on Eculizumab)
Number analyzed (Participants) | 10 | 8
score on a scale
  Week 1: number analyzed (Participants) | 9 | 8
  Week 1 | -0.2 (2.3) | 0.8 (1.8)
  Week 2: number analyzed (Participants) | 10 | 7
  Week 2 | 0.4 (2.2) | 0.1 (1.3)
  Week 3: number analyzed (Participants) | 10 | 7
  Week 3 | 0.3 (2.7) | 0.7 (1.8)
  Week 4: number analyzed (Participants) | 9 | 8
  Week 4 | -0.2 (2.0) | 0.4 (1.6)
  Week 6 | 0.3 (2.5) | 0.8 (2.3)
  Week 8 | -0.2 (2.3) | 0.3 (1.6)
  Week 10 | 0.3 (2.9) | 0.9 (1.6)
  Week 12: number analyzed (Participants) | 10 | 7
  Week 12 | -0.2 (2.9) | 0.0 (2.2)

ADVERSE EVENTS:
Time Frame: Through Week 12 of the study
Arm/Group | Cohort A (Treatment Naive) | Cohort B (Previously on Eculizumab)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/16
Serious Adverse Events (participants affected / at risk) | 2/10 | 1/16
Other Adverse Events (participants affected / at risk) | 10/10 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cohort A (Treatment Naive) (N=10) | Cohort B (Previously on Eculizumab) (N=16)
Pyrexia (General disorders) | 1 (1) | 0/0 (0) — General disorders and administration site conditions
Urinary tract Infection (Infections and infestations) | 0/0 (0) | 1 (1)
Febrile nonhaemolytic transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0/0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (Treatment Naive) (N=10) | Cohort B (Previously on Eculizumab) (N=16)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 1 (3)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 7 (7)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 3 (3)
Injection site bruising (General disorders) | 3 (3) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Crepitations (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Vaccination site pain (General disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Febrile nonhaemolytic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood glucose fluctuation (Investigations) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (3) | 7 (17)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (2) | 0 (0)
Device failure (Product Issues) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (2) | 0 (0)
Paroxysmal nocturnal haemoglobinuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure agreements are negotiated separately with each PI.

DOCUMENTS (2):
  • Study Protocol (2016-10-20): https://cdn.clinicaltrials.gov/large-docs/82/NCT03078582/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/82/NCT03078582/SAP_001.pdf